CLINICAL TRIAL: NCT04846140
Title: Identify Optimal Non-invasive Brain Stimulation Paradigm for Improving Peripheral Vision
Brief Title: Optimal Non-invasive Brain Stimulation for Peripheral Vision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); The University of Hong Kong (Other); University of Waterloo (Other); Hong Kong Metropolitan University (Other); Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Allen MY Cheong, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R5047-19
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma
Keywords: glaucoma; non-invasive brain stimulation; peripheral vision
MeSH Terms: conditions — Glaucoma | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 3 sessions of 3 types of active brain stimulation and 1 session of placebo sham stimulation. Each participant will perform four sessions in a randomly-assigned order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS group (Experimental): This group is defined as the participants who will receive tDCS at the first session. Participants in this group will receive 4 stimulation types (active a-tDCS, tACS, tRNS, and sham) in random order with at least a 48-hour separation between visits.
  Interventions: Device: transcranial electrical stimulation (tES)
- tACS group (Experimental): This group is defined as the participants who will receive tACS at the first session. Participants in this group will receive 4 stimulation types (active a-tDCS, tACS, tRNS, and sham) in random order with at least a 48-hour separation between visits.
  Interventions: Device: transcranial electrical stimulation (tES)
- tRNS group (Experimental): This group is defined as the participants who will receive tRNS at the first session. Participants in this group will receive 4 stimulation types (active a-tDCS, tACS, tRNS, and sham) in random order with at least a 48-hour separation between visits.
  Interventions: Device: transcranial electrical stimulation (tES)
- sham group (Experimental): This group is defined as the participants who will receive sham stimulation at the first session. Participants in this group will receive 4 stimulation types (active a-tDCS, tACS, tRNS, and sham) in random order with at least a 48-hour separation between visits.
  Interventions: Device: transcranial electrical stimulation (tES)

INTERVENTIONS:
Device: transcranial electrical stimulation (tES) — Transcranial electrical stimulation (tES) is a form of neuromodulation that uses constant, low direct current delivered via the electrodes on the skull. Three types of tES will be applied in this study, include a-tDCS, tACS, and tRNS. Additionally, sham stimulation will be applied as a placebo-controlled intervention.

SUMMARY:
Glaucoma is a complex disease that can result in progressive vision loss. There are no treatments that restore vision lost to glaucoma. However, recent studies have shown that vision can be improved by non-invasive brain (NIBS) stimulation and visual training. In this study, we aim to compare and find out the optimal non-invasive brain stimulation model (transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), and transcranial random noise stimulation (tRNS)) for improving peripheral vision in glaucoma patients. The proposed treatment is the application of transcranial electrical stimulation (tES) onto the participant's head, with brain stimulation aimed at the Primary Visual Cortex toward the occipital pole. The investigators hypothesize that the tES will enable higher performance in the reading task and secondary measures due to an increase in the cortical excitability of the stimulated brain cells, and tRNS will generate the greatest acute improvement in peripheral vision than either a-tDCS, tACS, or sham stimulation.

DETAILED DESCRIPTION:
This study uses a within-subjects, double-blind, placebo-controlled design and will be carried out in Hong Kong (The Hong Kong Polytechnic University).

Participants who will be recruited are 40 glaucoma patients aged 18 to 80, diagnosed with primary open-angle or normal-tension glaucoma with relative scotoma in both eyes. All participants will take part in 4 stimulation sessions (completion of active a-tDCS, tACS, tRNS, and sham stimulation in random order) with at least 48-hour separation between visits to wash out active stimulation effects.

The primary outcome is high-resolution perimetry that will be used to measure the visual field of participants. The secondary outcome is multifocal visual evoked potential (mfVEP) that will be used to measure the electrophysiological changes in the visual cortex.

The study consists of 5 visits:

Visit 1: Eligibility assessment (refer to the inclusion and exclusion criteria).

Visits 2 - 5: Stimulation sessions (completion of active a-tDCS, tACS, tRNS, and sham stimulation in random order) with at least 48-hours separation between visits to wash out active stimulation effects. An established protocol will be used. Briefly, active a-tDCS (2 mA), tACS (2 mA), tRNS (2 mA) or sham a-tDCS will be delivered for 20 minutes. The anodal electrode will be placed at Oz (visual cortex) while the cathodal electrode will be placed on the left cheek to facilitate stimulation of cells corresponding to the para-central retina that are located within the calcarine sulcus. Active stimulation will involve the delivery of 2 mA current continuously, while the fade-in-short-stimulation-fade-out approach will be used for the sham condition, in which the stimulation will be ramped down after 30 seconds of stimulation. Both the participant and experimenter will be masked to the stimulation type.

The average detection accuracy, response time, and functional connectivity will be analyzed using a within-subjects ANOVA with factors of Stimulation type (a-tDCS vs. tACS vs. tRNS vs. sham) and Time (pre and post-stimulation). Significant interactions will be investigated using post-hoc Bonferroni-adjusted paired sample t-tests. A significant interaction between Stimulation type and Time for the primary outcome followed by a significant post-hoc comparison with a p-value <0.05 favoring tRNS would be consistent with our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 80 years;
2. Diagnosis of primary open angle or normal tension glaucoma with relative scotoma in both eyes;
3. A relative scotoma defined as a Humphrey Field Analyser (HFA) threshold perimetry loss (mean deviation of ≤-6dB) within the central 30° of the visual field for at least one eye;
4. Best-corrected distance visual acuity of 6/12 or better (equivalent to 0.3 logMAR acuity or better to confirm that participant's central vision is preserved);
5. Stable vision and visual field loss for at least 3 months;
6. With a cognitive functional score of 22 or above in the Montreal Cognitive Assessment - Hong Kong version (HK-MoCA) (to confirm participant's intact cognitive function).

Exclusion Criteria:

1. Ocular diseases other than glaucoma (e.g. age-related macular degeneration, diabetic retinopathy, moderate to severe cataract) or severe hearing impairment (to ensure that participant can hear the instructions clearly during assessments and training);
2. Severe medical problems (e.g. stroke, Parkinson's disease) or self-reported neurological (e.g. brain surgery, brain tumor, peripheral neuropathy), or cognitive disorders (e.g. diagnosed dementia or cognitive impairment);
3. Self-reported vestibular or cerebellar dysfunction, history of vertigo;
4. Using any medications for any neurological conditions or psychiatric drugs (e.g. sedative, hypnotic) that might interfere with motor control;
5. Contraindications for non-invasive brain stimulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
High-resolution perimetry (HRP) | 0.5-1 hour
  Visual field will be measured using high-resolution perimetry (HRP, HighTechVision, Sweden), which is a valid and reliable computer-based campimetric visual field assessment. Suprathreshold stimuli will be presented in random order at 474 different positions to one eye (i.e. the eye with larger field loss) while fixation is monitored. Detection accuracy and response times will be recorded to map the patient's area of residual vision (i.e. relative scotoma). Testing will occur pre- and immediately post- stimulation.

SECONDARY OUTCOMES:
Multifocal visual evoked potential (mfVEP) | 0.5-1 hour
  Electrophysiological changes at visual cortex will be measured by multifocal visual evoked potential (mfVEP), a non-invasive neuroimaging technique related to electroencephalography (EEG) that is well established in the literature as a method for evaluating deficits in the visual field. Suprathreshold sectors of a circular checkerboard pattern will undergo visual reversal in a pseudorandom order to establish a visual evoked potential for each sector. Evoked potentials will be measured using a reference electrode placed at Fpz (i.e. forehead) and an array of 4 measurement electrodes arranged surrounding Oz (i.e. at the back of head). Subjects will be instructed to maintain fixation at the center of the screen while passively viewing the array of the stimulus, which will last approximately 12 minutes per session. Testing will occur pre- and immediately post- stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Cheong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Allen MY Cheong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be available upon reasonable request to the research team.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be available no later than 6 months following publication and for 1 year.
Access Criteria: IPD will be shared with investigators who provide a methodologically sound proposal.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT04846140/SAP_000.pdf